CLINICAL TRIAL: NCT03755973
Title: How do Different Ovarian Stimulation Protocols Affect Endometrial Receptivity During a Fresh In-vitro Fertilization Attempt
Brief Title: Effect of Different Ovarian Stimulation Protocols on Endometrial Receptivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidade de Lisboa (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1806-LIS-044-SD
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Infertility, Female; Endometrial Diseases
Keywords: Endometrial receptivity; Ovarian stimulation
MeSH Terms: conditions — Infertility, Female; Uterine Diseases | interventions — follitropin beta

STUDY DESIGN:
Intervention Model Description: All consenting subjects will first undergo an endometrial biopsy seven days after the luteinizing hormone (LH) peak in an unmedicated natural cycle. This biopsy will serve as the baseline endometrial biopsy (natural cycle biopsy) for the gene expression signature analysis. Following this baseline biopsy, the subjects will be randomly allocated to a specific type of ovarian stimulation regimen in order to later perform some second endometrial biopsy, five days after oocyte retrieval (stimulated cycle biopsy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CFA plus step-down rFSH (1A) (Experimental): A single dose of 150 IU of CFA followed by daily rFSH will be administered. The initial rFSH administration will be dosed between 100 IU and 200 IU according to the following criteria:
  * 200 or 300 IU: <3 follicles above 13 mm visible on transvaginal ultrasound;
  * 150 IU, >2 follicles above 13 mm and circulating day-8 follicle-stimulating hormone (FSH) levels ≤20 IU/mL.
  * 100 IU, >2 follicles above 13 mm and circulating day-8 FSH levels >20 IU/mL;
  Subjects will perform a step-down daily rFSH dose (fixed decreases in the dosing of 25 IU/day) until the triggering criteria are met or a minimum of 50 IU/day is reached. Subjects with <3 follicles above 13 mm visible will maintain 200 IU/day of rFSH until this criterion is met, initiating a fixed 25 IU/day stepdown protocol only from then onwards.
  Interventions: Drug: CFA; Drug: rFSH; Procedure: Step-down daily rFSH dose
- CFA plus fixed daily dose rFSH (1B) (Experimental): A single dose of 150 IU of CFA followed by a fixed daily rFSH dosing protocol of 200 or 300 IU will be administered as ovarian stimulation
  Interventions: Drug: CFA; Drug: rFSH; Procedure: Fixed daily rFSH dosing protocol of 200-300 IU
- Fixed daily dose rFSH only (Active Comparator): A fixed daily rFSH dosing protocol of 200 or 300 IU will be administered as ovarian stimulation
  Interventions: Drug: rFSH; Procedure: Fixed daily rFSH dosing protocol of 200-300 IU

INTERVENTIONS:
Drug: CFA — Long-acting exogenous ovarian stimulation
  Other Names: Corifollitropin alpha
  Arms: CFA plus fixed daily dose rFSH (1B); CFA plus step-down rFSH (1A)
Drug: rFSH — Daily rFSH
  Other Names: Puregon; Follitropin beta
Procedure: Fixed daily rFSH dosing protocol of 200-300 IU — The dose of daily rFSH is fixed at 200 or 300 IU
  Arms: CFA plus fixed daily dose rFSH (1B); Fixed daily dose rFSH only
Procedure: Step-down daily rFSH dose — The dose of daily rFSH is progressively reduced
  Arms: CFA plus step-down rFSH (1A)

SUMMARY:
This study will assess the change in endometrial gene expression signature on the day of embryo transfer according to the type of exogenous gonadotropins administered.

DETAILED DESCRIPTION:
Late-follicular elevated progesterone (LFEP) following ovarian stimulation for assisted reproductive technologies (ART) has been linked to abnormal endometrial receptivity expression profiles and lower pregnancy rates. For this reason, physicians frequently propose that patients with LFEP avoid performing a fresh embryo transfer, postponing instead it to a subsequent unstimulated cycle. Although this strategy may reduce the detrimental effect LFEP may have on cumulative ART pregnancy rates, it may also frustrate couples who wish to become pregnant as soon as possible.

With the intent of minimizing potentially-avoidable treatment delays, an increasing number of researchers are proposing that physicians revisit their current ovarian stimulation regimens. One strategy which may reduce the incidence of LFEP is to decrease the dose of gonadotropins administered at the end of stimulation (i.e. a stepdown protocol). A similar approach, using corifollitropin alpha (CFA), has also been recently advanced, taking advantage of the stepdown-like pharmacodynamic profile of this compound.

In order to assess the clinical usefulness of these strategies, the investigators propose a single-center, open-label, paired, randomized trial. The main objective of this study is to assess the changes in the endometrial gene expression profile on the day of fresh embryo transfer according to the type of gonadotropins administered for ovarian stimulation. In summary, all consenting subjects will first undergo an endometrial biopsy seven days after the luteinizing hormone peak in an unmedicated natural cycle. This biopsy will serve as the baseline endometrial biopsy (natural cycle biopsy) for a gene expression analysis. Following this baseline biopsy, subjects will be randomly allocated to a specific type of ovarian stimulation regimen in order to later perform a second endometrial biopsy, this time five days after oocyte retrieval (stimulated cycle biopsy). Subjects will be randomized to administer, on the third day of their menstrual cycle, either a single dose of 150 IU of CFA (study arms 1A and 1B) or a fixed daily dose of 200 or 300 IU of recombinant follicle stimulating (rFSH, study arm 2). On the eighth day of stimulation, it is expected that 15% to 30% of all subjects who performed CFA will have reached the follicular development criteria for final oocyte maturation and ovulation triggering.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form (ICF) dated and signed.
2. Age: ≥18 and ≤42 years old.
3. AFC <20.
4. AMH <2.5 ng/mL, performed in the 12 months prior to inclusion.
5. Body Mass Index (BMI): ≥18.5 Kg/m2 and <30 Kg/m2.
6. Weight: ≥50 kg and <80 kg.
7. First or second ART cycle (with pregnancy wish and planned for single blastocyst transfer) at the study site, or fertility preservation cycle.
8. Regular menstrual cycles (between 22 and 35 days).
9. Two ovaries present.

Exclusion Criteria:

1. Simultaneous participation in another clinical study.
2. Previous history of poor ovarian response (<4 oocytes retrieved) with a maximal dose of OS (≥300 IU/day) or OHSS, regardless of gonadotropin dose.
3. Known reasons for impaired implantation (i.e. hydrosalpinx, fibroid distorting the endometrial cavity, Asherman's syndrome, thrombophilia or endometrial tuberculosis).
4. Repeated miscarriages (>2 previous biochemical pregnancies or >2 spontaneous miscarriages).
5. Recurrent implantation failure (>3 failed cycles with good quality embryos).
6. Polycystic ovary syndrome (PCOS).
7. Tumours of the ovary, breast, uterus, pituitary or hypothalamus.
8. Abnormal (not menstrual) vaginal bleeding without a known/diagnosed cause.
9. Ovarian cysts or enlarged ovaries.
10. Fibroid tumours of the uterus incompatible with pregnancy.
11. Malformations of the reproductive organs incompatible with pregnancy.
12. Primary gonadal failure.
13. Renal impairment defined as estimated glomerular filtration rate of 90 ml/min/1.73 m2 determined by the Modified Diet and Renal Disease (MDRD) equation at screening.
14. Previous antibiotic hypersensitivity reactions (streptomycin and/or neomycin).
15. Risk factors for thromboembolic events, such as a personal or family history, severe obesity or thrombophilia.
16. Moderate or severe hepatic impairment.
17. Untreated and uncontrolled thyroid dysfunction.
18. Current use of oral contraceptive, anti-depressants, anti-psychotics, steroids, anti-epileptics or chemotherapy.
19. Administration of exogenous Estradiol (E2), Progesterone (P4) or gonadotropins in the preceding menstrual cycle.
20. Active female smoking.
21. Acceptors of donated oocytes/embryos.
22. Ongoing pregnancy.
23. Women who have previously enrolled in the trial.
24. Those unable to comprehend the investigational nature of the proposed study.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Endometrial gene expression signature on the day of embryo transfer | 7 days after the last day of ovarian stimulation
  RNA sequencing of specimen of endometrium

SECONDARY OUTCOMES:
Serum concentrations of progesterone from the start of stimulation until the day of embryo transfer | 3 weeks
  Measurement of serum circulating progesterone levels (in ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Santos-Ribeiro, MD PhD, Principal Investigator — Instutito Valenciano de Infertilidade de Lisboa
Locations (1):
- Instituto Valenciano de Infertilidade, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No